CLINICAL TRIAL: NCT04844281
Title: Evaluation of Wear Experience With PRECISION1® Toric Contact Lenses on Long Lens Wear Days
Brief Title: Wear Experience With Daily Toric Contact Lenses Over a Long Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Associate Professor of Clinical Optometry, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0559
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Contact Lens; Astigmatism of Both Eyes
Keywords: Toric Contact Lens; Daily Contact Lens

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Daily Disposable Toric Contact Lens (Experimental): All subjects are fit into Precision1® toric contact lenses. Subjects are requested to wear the lenses for a total of two weeks.
  Interventions: Device: Precision1® Daily Disposable Toric Contact Lens

INTERVENTIONS:
Device: Precision1® Daily Disposable Toric Contact Lens — Soft, toric contact lens used to correct distance vision and astigmatism.

SUMMARY:
This study is evaluating the wear experience of a daily toric contact lens after 10, 12, 14, and 16 hours of lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Must be current soft toric contact lens wearers with longs days of lens wear within the parameters of Precision1® lenses available.
* Distance visual acuity of 20/25 or better with current lenses.
* Recent eye exam in the last year.
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI).
* Ability to give informed consent.
* Must have a working smart phone or device and be willing to receive and respond to texts and/or emails.
* Willing to spend time for the study, which includes three in-person study visits (with a possible fourth visit if needed), wearing contact lenses on days between study visits, and responding to communications on a smart phone or other electronic device on five weekdays between Visits 2 and 3.

Exclusion Criteria:

* Current ocular inflammation or infection as assessed by the study investigator.
* Currently pregnant, lactating, or planning to become pregnant during the course of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Disposable Toric Contact Lens
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daily Disposable Toric Contact Lens
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Subjective Vision in Contact Lenses Assessed Using a 1 to 10 Scale After 16 Hours of Wear in One Day (After up to 14 Days of Wear)
Description: 1 describes poor experience, and 10 describes excellent experience.
Time Frame: Assessment is taken at the 16 hour of wear time point in a single day, after up to 14 days of wear.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Daily Disposable Toric Contact Lens
Number analyzed (Participants) | 30
units on a scale | 9 [7 to 10]

2. Primary Outcome: Subjective Comfort on a 1-10 Scale After 16 Hours of Wear in One Day (After up to 14 Days of Wear)
Description: 1 describes poor experience, and 10 describes excellent experience.
Time Frame: Taken at the 16 hour of wear time point in a single day, after up to 14 days of wear Up to 14 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Daily Disposable Toric Contact Lens
Number analyzed (Participants) | 30
units on a scale | 8.4 [7 to 9]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Daily Disposable Toric Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04844281/Prot_002.pdf